CLINICAL TRIAL: NCT04255641
Title: Is Morphokinetic Scoring by Time - Lapse Analysis of Embryos Undergoing Cryopreservation During IVF Associated With Post- Thaw Survival and Treatment Outcome: A Retrospective Analysis
Brief Title: Time - Lapse Analysis of Frozen Embryos
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMC-19-0121-CTIL
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Frozen Embryos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- frozen embryos
  Interventions: Other: time lapse analysis

INTERVENTIONS:
Other: time lapse analysis — grading of the embryos before freezing using time lapse/

SUMMARY:
A retrospective analysis of embryo defrost cycles that were rated in the EmbryoScope system and frozen will be performed. The study will examine the possible association between the morphokinetic grading received by these embryos as fresh embryos before freezing, and their survival, the morphological grading they received after thawing, their proper rooting and live birth after thawing.

ELIGIBILITY:
Inclusion Criteria:

* All women who underwent embryo freezing and thawing between the years 2014-2019 in Carmel medical center

Exclusion Criteria:

* Lack of proper data

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All women who underwent embryo freezing and thawing between the years 2014-2019 in Carmel medical center
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
live birth | 1 day
embryos survival after thawing | 1-2 days
implantation in the uterus | 1 week
post thaw grading | 1 day
  post thaw grading of the embryos using time lapse analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided